CLINICAL TRIAL: NCT02005003
Title: Placebo-controlled Randomized Trial of Cognitive and Metabolic Effects of a Probiotic Supplement
Brief Title: Cognitive and Metabolic Effects of a Probiotic Supplement
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Uppsala University (Other)
Responsible Party: Principal Investigator, Jonathan Cedernaes, Medical doctor, PhD, Uppsala University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: FF8vsPlaceboJC2013
Record Dates: First submitted 2013-11-27; First posted 2013-12-09 (Estimated); Last update posted 2014-11-18 (Estimated); Status verified 2014-11

CONDITIONS: Dietary Supplements; Probiotics; Metabolism; Food Preferences; Microbiota
MeSH Terms: conditions — Food Preferences | interventions — Blood Specimen Collection

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Probiotic (Active Comparator): Probiotic pills given for 2 weeks, during one of the interventions that the participants is either randomized to as the first or second intervention period. At day 0 and following each intervention period (at week 2 and week 6), participants will be tested using Inhibitory task, Blood samples, Feces collection, Caloric preload, Food selection task, Memory task and Food consumption task.
  Interventions: Behavioral: Inhibitory task; Procedure: Blood samples; Biological: Feces collection; Procedure: Caloric preload; Behavioral: Food selection task; Behavioral: Memory task; Behavioral: Food consumption task
- Placebo (Placebo Comparator): Placebo pills given for 2 weeks, during one of the interventions that the participants is either randomized to as the first or second intervention period. At day 0 and following each intervention period (at week 2 and week 6), participants will be tested using Inhibitory task, Blood samples, Feces collection, Caloric preload, Food selection task, Memory task and Food consumption task.
  Interventions: Behavioral: Inhibitory task; Procedure: Blood samples; Biological: Feces collection; Procedure: Caloric preload; Behavioral: Food selection task; Behavioral: Memory task; Behavioral: Food consumption task

INTERVENTIONS:
Behavioral: Inhibitory task — Participants perform a binary decision on each presented stimuli. Of the two possible outcomes, participants are instructed to make a motor response (go) for one type, and are to withhold a response (no-go) for the other type. Reaction time and accuracy are measured for each event
Procedure: Blood samples — Hormone levels will be analyzed from blood samples obtained before and after a caloric preload given at each visit
Biological: Feces collection — Feces samples will be collected on the morning of each visit, before and after each 2-week intervention period, as well as after each 2-week washout period following each intervention period.
Procedure: Caloric preload — A caloric preload will be given to participants, following which blood will be taken at 65 minutes later (specified in Blood sampling) following the ingestion of the caloric preload.
Behavioral: Food selection task — Participants are given the opportunity to write and use a computer program to specify amount and type of food would ideally like to consume
Behavioral: Memory task — Participants perform short memory tasks on each visit
Behavioral: Food consumption task — Participants are given a selection of food items to consume on each visit

SUMMARY:
To examine the cognitive and metabolic effects of a probiotic supplement that is readily and already available for purchase in public drug stores. This study is a double-blinded randomized cross-over placebo-controlled intervention study. Participants will be randomized to receive either the probiotic supplement or the placebo during the first intervention period which will last 2 weeks. This will be followed by a washout period, after which they will proceed to the second intervention period, also lasting 2 weeks and also followed by a washout period.

ELIGIBILITY:
Inclusion Criteria:

* Male
* Age 18-28y
* Healthy (self-reported) and not on medication
* Non-smoking
* Normal sleep-wake rhythm (i.e. 7-8 h per night, self-reported via diaries)
* Regular meal patterns with daily breakfast

Exclusion Criteria:

* Major illness
* Taking any serious medications
* Any sleep conditions (e.g. irregular bedtimes, sleep complaints)
* Any dietary issues with the food items provided
* Current or history of endocrine, neurological or psychiatric disorders
* Shift work in the preceding three months or for a long duration
* Time travel over a significant number of time zones in the preceding two months
* Too much weight gain or weight loss in the preceding three months
* Excessive intake of fermented dairy products
* Intake of probiotics
* Recent antibiotic treatment (last 6 months)
* Recent intake of certain dietary supplements
* Excessive caffeine (>5 cups daily) or alcohol intake (>2 alcohol units daily)

Ages: 18 Years to 28 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2013-11; Primary Completion 2015-12 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Memory function | Change in memory function assessed at baseline (week 0), post-intervention 1 (at week 2), pre intervention 2 (week 6), post intervention 2 (week 8) and post-washout intervention 2 (week 12)
  Memory test to examine the influence of probiotic supplement compared with placebo on memory function (declarative and working memory)

SECONDARY OUTCOMES:
Glycometabolic regulation | Change in glycometabolic regulation assessed at baseline (week 0), post-intervention 1 (at week 2), pre intervention 2 (week 6), post intervention 2 (week 8) and post-washout intervention 2 (week 12)
  Glucose, insulin and other hormonal values during fasting and 1 hour following a standardized caloric preload
Food preferences | Change in food preferences assessed at baseline (week 0), post-intervention 1 (at week 2), pre intervention 2 (week 6), post intervention 2 (week 8) and post-washout intervention 2 (week 12)
  Will test whether participants food preferences are changed following each intervention, as compared with before each intervention. Test will be written and computer-based.
Inhibitory task | Change in inhibitory task performance assessed at baseline (week 0), post-intervention 1 (at week 2), pre intervention 2 (week 6), post intervention 2 (week 8) and post-washout intervention 2 (week 12)
  Participants perform a binary decision on each presented stimuli. Of the two possible outcomes, participants are instructed to make a motor response (go) for one type, and are to withhold a response (no-go) for the other type. Reaction time and accuracy are measured for each event.
Food consumption task | Change in food consumption task assessed at baseline (week 0), post-intervention 1 (at week 2), pre intervention 2 (week 6), post intervention 2 (week 8) and post-washout intervention 2 (week 12)
  Participants will be offered a food selection and their consumption will be measured.
Sleep patterns | Change in sleep patterns as assessed at baseline (week 0), post-intervention 1 (at week 2), pre intervention 2 (week 6), post intervention 2 (week 8) and post-washout intervention 2 (week 12)
Microbiome changes | Microbiome assessed at baseline (week 0), post-intervention 1 (at week 2), pre intervention 2 (week 6), post intervention 2 (week 8) and post-washout intervention 2 (week 12)
  Changes in microbiome will be assessed following treatment with either placebo or probiotics; feces will be collected according to standardized criteria.

CONTACTS AND LOCATIONS:
Overall Officials: Christian Benedict, PhD, Principal Investigator — Department of Neuroscience, Uppsala University
Locations (1):
- Department of Neuroscience, Uppsala University, Uppsala, Sweden